CLINICAL TRIAL: NCT02266836
Title: Clinical Feasibility and Usability of MyndMove Therapy for FES Facilitated Treatment of Subacute and Chronic Severe Hemiparesis of the Upper Limb Following Stroke
Brief Title: MyndMove Therapy for Severe Hemiparesis of the Upper Limb Following Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MyndTec Inc. (Industry)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT-ST-2001
Record Dates: First submitted 2014-09-26; First posted 2014-10-17 (Estimated); Last update posted 2020-01-28 (Actual); Status verified 2019-08

CONDITIONS: Hemiparesis of the Upper Limb Following Stroke
Keywords: Stroke; Cerebrovascular accident; Upper Extremity; Cerebral Infarction; Brain Infarction; Brain Ischemia; Cerebrovascular Disorders; Cardiovascular Diseases; Nervous System Diseases; Central Nervous System Diseases
MeSH Terms: conditions — Stroke; Cerebral Infarction; Brain Infarction; Brain Ischemia; Cerebrovascular Disorders; Cardiovascular Diseases; Nervous System Diseases; Central Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MyndMove (Experimental): The MyndMove system is a neuromodulation device that delivers short electrical pulses to stimulate muscle contractions and enhance motor recovery following Stroke or Spinal Cord Injury. MyndMove delivers therapeutic stimulation sequences called protocols, which are coded therapeutic algorithms which assist muscle movement allowing the brain and central nervous system to be retrained restoring voluntary reaching and grasping functions lost following neurological injury. The MyndMove system comprises the hardware device, stimulation electrodes and cables, hand and foot switches, and integrated software.
  Interventions: Device: MyndMove

INTERVENTIONS:
Device: MyndMove — During a MyndMove therapy session, the patient is instructed to attempt to execute a task voluntarily. As the patient is attempting to perform the designated task, specific muscles in the arm are stimulated to generate contractions that produce the desired movement. After a brief interval of the patient attempting to initiate a movement the therapist activates the MyndMove stimulation protocol, which generates bursts of short electrical pulses, using surface electrodes, to produce muscle contractions enabling the patient to complete the desired/instructed task. Proper sequencing of the muscle contractions as per the MyndMove protocols are tailored to achieve a wide range of reaching and grasping functions. The technique stimulates non-damaged pathways of the central nervous system.

SUMMARY:
The purpose of this study is to examine the efficacy of MyndMove therapy in the early sub-acute, late sub-acute and chronic post-stroke patients. Other objectives include assessing the required doses of electrical current amplitudes, the usability of the device, and examining the overall safety.

DETAILED DESCRIPTION:
The purpose of this study is to examine the efficacy of MyndMove therapy in the early sub-acute, late sub-acute and chronic post-stroke patients. Other objectives include assessing the required doses of electrical current amplitudes, the usability of the device, and examining the overall safety.

Many individuals experience weakness or paralysis of their arms and hands following a stroke. As a result, they are often unable to grasp and reach objects voluntarily and have difficulty performing basic activities of daily living (ADLs) such as dressing, feeding, bathing and grooming. Despite extensive rehabilitation programs, many of these individuals remain dependent on others for assistance with ADLs. This unmet medical need remains the focus of a wide range of research efforts.

MyndMove is a newly developed Functional Electrical Stimulation based treatment designed to recover voluntary movement in severely paralyzed upper limbs following stroke and spinal cord injury.

This study will enroll stroke patients that have severe hemiparesis of an upper limb (as defined by 1) an UE-FMA score of less than or equal to 19 and 2) a Chedoke McMaster Stage of 1-2 for the arm and hand). Three cohorts of patients enrolled in the study will include:

* Early sub-acute stroke patients (less than 2 months post stroke) receiving therapy during inpatient rehabilitation;
* Late sub-acute stroke patients (post-discharge from inpatient rehab and less than 6 months post stroke) receiving therapy in outpatient clinic settings; and
* Chronic stroke patients (greater than 6 months post stroke) receiving therapy in outpatient clinic settings

ELIGIBILITY:
Inclusion Criteria:

1. Ischemic or hemorrhagic stroke confirmed by MRI or CT scan
2. Sub-acute subjects at least 10 days post stroke. Chronic subjects at least 6 months post stroke
3. Chedoke-McMaster Stroke Assessment Stage 1-2 (arm and hand)
4. Severe hemiplegia of the upper extremity defined as UE-FMA score of less than or equal to 19
5. Subject is able to follow instructions
6. Subject is able to sit and participate in one hour of upper limb therapy
7. Anticipated to be discharged home or already at home following conventional inpatient rehabilitation
8. Willing to attend outpatient therapy if chronic or late sub-acute
9. Subject is able and willing to give written informed consent
10. Men and women aged 18 or older

Exclusion Criteria:

1. Global Aphasia
2. Previous history of clinical stroke either ischemic infarct, hemorrhagic and subarachnoid bleeding
3. Upper extremity injury or condition prior to stroke that limits the function of the hand or arm
4. Life expectancy of less than 12 months due to other illness
5. Subject has malignant skin lesion on the affected upper extremity
6. Subject has history of seizure disorder and on seizure medications
7. Subject has existing electrical stimulation devices (ICD, Pacemaker, Spinal Stimulation)
8. Neurologic condition that may affect motor response (e.g. Parkinson's, ALS, MS)
9. Subject has rash or open wound at any potential electrode site
10. In the judgment of the medical provider, subject has medical complications that may interfere with the execution of the study
11. Botulinum toxin (Botox) injection into affected upper extremity at least 3 months before the study or during the study
12. Currently enrolled in another upper limb study
13. Enrolled in the past six months in a clinical study involving drugs or biologics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in Upper Extremity Fugl-Meyer Assessment (UE-FMA) | baseline to 6 weeks
  The Upper Extremity Fugl-Meyer Assessment (UE-FMA) is a standardized scale used for the evaluation of physical performance in the post-stroke hemiplegic patient. The upper extremity (UE) evaluates the function of the upper extremity motor function in four components: Shoulder/Elbow and Forearm, Wrist, Hand and Coordination and Speed in a series of performed tasks. The maximum score associated with the UE-FMA is 66 points. Each of the 33 specific tasks is scored as either 0 or an absence of function to a maximum score of 2 for the tasks being fully completed. Partial function can be scored as 1 for selected tasks. This evaluation will be completed by a trained physiotherapist or occupational therapist. Upper extremity assessment for stroke patients. Clinically Significant change is >6 points

SECONDARY OUTCOMES:
Change in Functional Independence Measure and Self-Care Functional Independence Measure for the early subacute subjects | Baseline - 6 weeks
  To measure the degree of disability the Functional Independence Measure will be completed. The FIM consists of 18 items of which 13 are motor related tasks and 5 are cognitive related items. The measure is broken down into 6 classifications of self-care, sphincter control, mobility, locomotion, communication and social cognition. The self-care consists of 6 items: eating, grooming, bathing, dressing-upper body, dressing-lower body, toileting. Each item is rated using a 7-point scale indicating the level of functioning from total assistance with a score of 1 to complete independence with a score of 7.
System Usability Scale | An average of 5 weeks after therapy has begun
  Each Therapist will complete the System Usability Scale on the last treatment visit which is expected to be an average of 5 weeks after therapy has begun. Each question in the System Usability Scale is scored from 1 - Strongly Disagree, through to 5 - Strongly Agree. System Usability Scale scores, based on therapist assessments, at end of study compared to baseline (after basic training).
All adverse events | Baseline - An average of 5 weeks after therapy has begun
  At each study visit, participants will be asked if they have experienced any adverse events. Participants will be in the study for an expected average of 5 weeks.
Amplitudes to elicit muscle movement | Throughout study
  The amplitudes that are used to elicit the muscle movement will be recorded for the various muscles for each participant. The average required amplitude will be calculated and the minimum and maximum amplitudes will be noted. This will provide future guidance on the typical range of amplitudes needed for the various muscles to treat patients.

CONTACTS AND LOCATIONS:
Overall Officials: Debbie A Hebert, MSc(Kin), Principal Investigator — University Health Network, Toronto; Mark Bayley, MD, Principal Investigator — University Health Network, Toronto
Locations (6):
- Canada (6):
  - Brampton, Ontario
  - London, Ontario
  - Oshawa, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Windsor, Ontario